CLINICAL TRIAL: NCT02084004
Title: Effects of Berberine Hydrochloride and Bifidobacterium in Diabetes Mellitus Prevention and Treatment：an Open-label, Multicenter，Randomized, Prospective，Controlled Study
Brief Title: Effects of Berberine Hydrochloride and Bifidobacterium in Diabetes Mellitus Prevention and Treatment
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: The sponsor have not enough money to support this trial
Sponsor: Xijing Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2013KTZB03-02-01A
Record Dates: First submitted 2014-02-27; First posted 2014-03-11 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Type 2 Diabetes Mellitus
Keywords: Type 2 diabetes mellitus; Berberine Hydrochloride; Bifidobacterium
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Bifidobacterium viable pharmaceutics (Experimental): Bifidobacterium viable pharmaceutics, 2 Capsules, 2/day, 12 weeks
  Interventions: Drug: Bifidobacterium viable pharmaceutics
- Berberine Hydrochloride (Experimental): Berberine Hydrochloride, 0.5g, 2/day, 12 weeks
  Interventions: Drug: Berberine Hydrochloride
- lifestyle counseling (No Intervention)

INTERVENTIONS:
Drug: Bifidobacterium viable pharmaceutics
  Arms: Bifidobacterium viable pharmaceutics
Drug: Berberine Hydrochloride
  Arms: Berberine Hydrochloride

SUMMARY:
The aim of this study is to assess the beneficial effects of Bifidobacterium Hydrochloride and Berberine on lowering glucose in patients with type 2 diabetes mellitus and to detect the potential mechanism.

DETAILED DESCRIPTION:
Gut microbiota maybe play an important role in patients with type 2 diabetes mellitus (T2DM). Berberine, which is usually used as an antibiotic drug, has been reported a potential glucose-lowering effect in vitro and in vivo studies. Bifidobacterium, as a familiar probiotics, can modulate gut microbiota and improve glucose and lipid metabolism in animal experiments. Therefore, the aim of this study is to assess the beneficial effects of Bifidobacterium Hydrochloride and Berberine on lowering glucose in patients with T2DM and to detect the potential mechanism.

ELIGIBILITY:
Inclusion Criteria:

* Informed consent obtained before any trial-related activities；
* Male or female between 18 and 70 years of age
* 19≤Body mass index(BMI)≤30kg/m2
* No participate in any clinical trial at least 3 months
* Newly diagnosed T2DM (OGTT) or not received previous pharmacological treatment
* 7%≤HbA1c≤9%
* Females in child-bearing period should be given birth control
* No severe disease about heart, lung and kidney
* Ability and willingness to adhere to the protocol including performance of self-monitored blood glucose (SMBG) profiles according to the protocol
* Subject is likely to comply with the Investigators instruction

Exclusion Criteria:

* Type 2 or 1 diabetes mellitus received previous pharmacological treatment
* Females of childbearing potential who are pregnant，breastfeeding or intend to become pregnant or are not using adequate contraceptive methods
* Impaired liver function, defined as Aspartate aminotransferase（AST） or Alanine transaminase (ALT)> 2 times upper limit of normal (central laboratory)
* Impaired renal function, defined as serum-creatinine≥133μmol/L
* Uncontrolled treated/untreated severe hypertension (systolic blood pressure≥160mmHg and /or diastolic blood pressure≥95mmHg)
* Chronic gastrointestinal diseases
* Cancer and medical history of cancer (except basal cell skin cancer or squamous cell skin cancer)
* Any clinically significant disease or disorder, which in the Investigator's opinion could interfere with the results of the trial
* Mental incapacity, psychiatric disorder, unwillingness or language barriers precluding adequate understanding or co-operation, including subjects not able to read and write
* Previous participation in this trial. Participation is defined as randomized. Re-screening of screening failures is allowed only once within the limits of the recruitment period
* Known or suspected hypersensitivity to trial products or related products
* Known or suspected abuse of alcohol, narcotics or illicit drugs

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-11 (Estimated); Primary Completion 2018-04 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Change in HbA1c from baseline to week 12 | Baseline and week 12
  Change was measured at baseline and week 12 after randomization. Change was reported as the absolute difference in % HbA1c.

SECONDARY OUTCOMES:
Percentage of subjects achieving HbA1c < 7% at week 12 | Week 12
Gut microbiome composition | Baseline and week 12
  Faecal bacterial composition determined from microbiological cultures and deep metagenomic next-generation sequencing of bacterial DNA in feces.
Changes in postprandial glucagon-like peptide-1 (GLP-1) secretion between baseline and week 12 | Baseline and week 12
  Plasma level of GLP-1 at baseline and week 12 during a 2 hour-meal test.
Adverse effects | From baseline to week 12
  Standardized questionaries regarding gastrointestinal function are filled out at each study visit (0, 4, 8 and 12 weeks after randomization) to detect possible adverse effects of antibiotics. In addition, subjects are given a calendar and informed to write down any symptom or illness during the study period.

CONTACTS AND LOCATIONS:
Overall Officials: Qiuhe Ji, Ph.D.,M.D., Principal Investigator — Department of Endocrinology, Xijing Hospital, Fourth Military Medical University
Locations (4):
- China (4):
  - Second Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - The 323rd Hospital of People's Liberation Army, Xi'an, Shaanxi
  - First Affiliated Hospital of Xi'an Jiaotong University, Xi'an, Shaanxi
  - Shaanxi Provincial People's Hospital, Xi'an, Shaanxi